CLINICAL TRIAL: NCT01048580
Title: A Phase I Study of Perifosine + Capecitabine for Patients With Advanced Colon Cancer
Brief Title: Study of Perifosine + Capecitabine for Colon Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 141
Record Dates: First submitted 2010-01-09; First posted 2010-01-13 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2011-11

CONDITIONS: Colon Cancer
Keywords: Perifosine; Capecitabine; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — perifosine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perifosine +Capecitabine (Experimental): One cycle of therapy will be defined as 3 weeks (21 days). Perifosine 50 mg qd (Days 1-21) + Capecitabine 1000 mg/m2 BID (Days 1-14).
  Interventions: Drug: Perifosine; Drug: Capecitabine

INTERVENTIONS:
Drug: Perifosine — Perifosine 50 mg orally once a day (Days 1-21)
  Other Names: D-21266; KRX-0401
Drug: Capecitabine — Capecitabine 1000 mg/m2 orally twice per day (Days 1-14)
  Other Names: Xeloda

SUMMARY:
This is a Phase I study of Perifosine + Capecitabine for patients with advanced colon cancer.

DETAILED DESCRIPTION:
This study is a Phase I trial. A total of 3 - 9 patients will be enrolled. Three patients will initially be enrolled. There will be no dose escalation in this study as only one dose for perifosine (50 mg) in combination with one dose of capecitabine (1000 mg/m2 BID) will be evaluated. The maximum tolerated dose (MTD) is defined in which fewer than 33% of patients experienced DLT attributable to the study drug(s), when at least six patients have been treated at that dose and are evaluable for toxicity. Pharmacokinetic (PK) data will also be evaluated from all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 3rd line or > metastatic colon cancer
* Patients must have received or not be candidates for regimens containing 5- FU, oxaliplatin, irinotecan, bevacizumab, and cetuximab or panitumumab
* No prior exposure to perifosine
* Adequate bone marrow, liver, and renal function
* Patients must have at least one measurable lesion
* Patients must agree to have extra blood drawn for PK analyses

Exclusion Criteria:

* Patients with prior exposure to perifosine.
* Patients receiving any other investigational agents or devices.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* Patients with known dipyrimidine dehydrogenase (DPD) deficiency or prior severe reaction to 5-FU.
* Patients with known central nervous system CNS metastases.
* Patients with known HIV, Hepatitis B, or Hepatitis C seropositivity.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), or New York Heart Association class II-IV congestive heart failure.
* Female patients who are pregnant or lactating are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the combination of perifosine and capecitabine (i.e., dose limiting toxicity) | Every 3 weeks after dosing
  The maximum tolerated dose (MTD) is defined in which fewer than 33% of patients experienced dose limiting toxicity (DLT) attributable to the study drug(s), when at least six patients were treated at that dose and are evaluable for toxicity. A DLT will be defined as any of the following deemed to be related to study drug(s):
  * Grade 3 non-hematologic toxicity except alopecia not reversible to Grade 2 or less within 96 hours
  * Any Grade 4 toxicity DLT will be based on the first cycle of treatment (first 21 days). Toxicity will be graded according to the NCI CTCAE version 3.0. To be evaluable for toxicity, a patient must receive at least 1 complete course of treatment or have experienced DLT.

SECONDARY OUTCOMES:
Best overall response | Every 3 cycles after dosing (length of one cycle is 21 days)
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  Response Evaluation Criteria in solid tumors (RECIST): Measurable disease is defined as the presence of at least one measurable lesion. Measurable lesions are lesions that can be accurately measured in at least one dimension and fit one of the following criteria:
  1. Longest diameter ≥ 20 mm using conventional techniques, or
  2. ≥ 10 mm with spiral CT scan.
Time to progression | Every 3 cycles after dosing (length of one cycle is 21 days)
  This is the interval from the initiation of treatment to the time of documented, objective progression using the same methods of evaluation that were used at baseline.
  In order for a patient to be regarded as having progressive disease, the following criteria must be met:
  1. The site of disease must have been evaluated either at baseline or while receiving study medication. Both evaluations must use the same methodology.
  2. PET scan results will not be used as evidence of either progression or response..
Pharmacokinetic (PK) data for the combination of perifosine and capecitabine | Up to cyle 5 no pharmacokinetic samples were obtained. Cycle 1/Day 11 until Cycle 4/Day 11: pharmacokinetic samples obtained 0.5, 1, 2, 4, 6 and 8 hours after dosing
  PK data will also be evaluated from all enrolled patients. PK analyses will present peak plasma concentrations (Cmax) as well as Area under the plasma concentration verus time curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell,, MD, Study Chair — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Journal of Oncology, 2010 ASCO Annual Meeting Abstracts. Vol. 28, No. 15_suppl (May 20Supplement), 2010:e14086